CLINICAL TRIAL: NCT04436965
Title: Effect of Standard Nutrition Therapy on Nutritional Status and Prognosis in Locoregionally Advanced Nasopharyngeal Carcinoma Patients With Malnutrition: A Prospective, Multicenter, Phase III Randomized Control Clinical Trial
Brief Title: Effect of Standard Nutrition Therapy on Nutritional Status and Prognosis in Locoregionally Advanced Nasopharyngeal Carcinoma Patients With Malnutrition
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wuhan University (Other); The First Affiliated Hospital of Xiamen University (Other); Fudan University (Other); Jiangxi Provincial Cancer Hospital (Other); Xijing Hospital (Other); Xiangya Hospital of Central South University (Other); Fujian Cancer Hospital (Other Government); Zhejiang Cancer Hospital (Other); Cancer Hospital of Guizhou Province (Other)
Responsible Party: Principal Investigator, Zhao Chong, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-FXY-348-NPC
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Nasopharyngeal Carcinoma; Nutrition Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard nutrition therapy (Experimental): Dynamic nutrition assessment will be performed to patients. If malnutrion happened, patients would receive oral nutritional supplements (ONS) first, then feeded with nasal feeding tube or PEG when ONS wasn't enough. If all the these enteral nutrition methods couldn't make up for patient's nutritional deficiencies, parenteral nutrition would be considered.
  Interventions: Other: Standardized nutrition therapy; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy
- Conventional nutrition therapy (Active Comparator): Dynamic nutrition assessment will be performed to patients throughout whole treatment, and symptomatic treatment would be performed if needed.
  Interventions: Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Other: Standardized nutrition therapy — Standardized nutrition therapy with ONS, nasal feeding tube, PEG or parenteral nutrition
  Arms: Standard nutrition therapy
Drug: Cisplatin — Patients in both arms received concurrent cisplatin chemotherapy:100 mg/m² cisplatin given intravenously every 3 weeks on days 1, 22 concurrently with radiotherapy.
  Other Names: DDP
Radiation: Intensity Modulated Radiation Therapy — Patients in both arms received Intensity Modulated Radiation Therapy:All target volumes were outlined slice by slice on the axial contrast-enhanced CT with MR fusion images in the treatment planning system. The target volumes were defined in accordance with the International Commission on Radiation Units and Measurements Reports 83. The prescribed dose was 70-72 Gy to PTVnx (Planning target volume of the primary tumor), 64-70 Gy to PTVnd (Planning target volume of the cervical lymph node),60- 64Gy to PTV1 (Planning target volume 1), and 54-58 Gy to PTV2 (Planning target volume 2) in 30-32 fractions. The details of dose limits for organs at risk were based on the study 0225 from The Radiation Therapy Oncology Group (RTOG 0225).
  Other Names: IMRT

SUMMARY:
This is a multicenter, randomized controlled, phase III clinical trial. The purpose of this study is to evaluate the efficacy of standard nutrition treatment versus conventional nutrition treatment in local advanced nasopharyngeal carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma(WHO II/III);
* All genders，range from 18～65 years old;
* Karnofsky performance status(KPS) ≥ 80;
* Clinical stage III~IVa(AJCC/UICC 8th);
* Without significant digestive system disease，nutritional and metabolic diseases or endocrine disease
* Without significant cardiac，respiratory，kidney or liver disease;
* Not received radiotherapy, chemotherapy and other anti-tumor treatment(including immunotherapy);
* White blood cell(WBC) count ≥ 4×109/L, neutrophile granulocyte(NE) count ≥ 1.5×109/L, Hemoglobin(HGB) ≥ 9g/L, platelet(PLT) count ≥ 100×109/L
* Total bilirubin(TBIL)、alanine aminotransferase (ALT) or aspartate aminotransferase(AST) < 2.5×upper limit of normal(ULN);
* Adequate renal function: BUN/CRE ≤ 1.5×ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* No contraindications to chemotherapy or radiotherapy;
* Inform consent form;

Exclusion Criteria:

* Have some PEG/PEJ contraindications, such as coagulopathy, recent anticoagulant medications and aspirin, gastric ulcer or history of gastric bleeding, portal hypertension combined with abdominal and esophageal fundal varices, pyloric obstruction due to residual stomach under the costal arch after various major gastrectomy or various reasons;
* Distance metastases;
* Have or are suffering from other malignant tumors;
* Participating in other clinical trials;
* Drug or alcohol addition;
* Do not have full capacity for civil acts;
* Mental disorder;
* Pregnancy or lactation;
* Severe complication, eg, uncontrolled hypertension;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of IBW% | 2 months
  To observe the changes and differences in the incidence of the actual weight/ideal weight (IBW%) less than 90% during the treatment of the two groups of patients

SECONDARY OUTCOMES:
The incidence of WL、UBW% and BMI | 36 months
  To observe the changes and differences in the incidence of body weight loss (WL)≥5%/10%, actual body weight/usual body weight (UBW%), body mass index (BMI) before, during and after treatment
Number of Participants With Abnormal Laboratory Values | 36 months
  To observe patients' complete blood cell count and blood biochemical examination during the treatment and three years after the treatment.
Overall survival | 36 months
  From date of recruited to death
Progression free survival | 36 months
  From date of recruited to disease progression
Locoregional recurrence free survival | 36 months
  From date of recruited to locoregional recurrence
Distant metastasis free survival | 36 months
  From date of recruited to distant metastasis
Nutrition screening and evaluation | 36 months
  To observe the changes and differences of nutrition screening and evaluation (NRS2002 and PG-SGA) before, during and after treatment in the two groups
Quality of life: EuroQoL 5 dimension | 36 months
  Evaluating with questionnaire of EuroQoL 5 dimension, 5 level health state utility index (EQ-5D-5L)
Acute toxicities | through study completion, an average of 2 months
  Evaluating with CTCAE v5.0
Late toxicity | 36 months
  assessed with Radiation Therapy Oncology Group radiation morbidity scoring criteria

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn